CLINICAL TRIAL: NCT01027598
Title: A Randomized Phase II Double-Blind Trial of Erlotinib and Pazopanib, or Erlotinib and Placebo in Patients With Previously Treated Advanced Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Randomized, Double-Blind Trial of Erlotinib/Pazopanib or Erlotinib/Placebo in Patients With Previously Treated Advanced Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCRI LUN 200
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer; Previously Treated Advanced Non Small Cell Lung Cancer; Erlotinib; Pazopanib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pazopanib; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib + Pazopanib (Experimental): Erlotinib: 150 mg orally daily
  Pazopanib: 600 mg orally daily
  Interventions: Drug: Pazopanib; Drug: Erlotinib
- Erlotinib + Placebo (Placebo Comparator): Erlotinib: 150 mg orally daily
  Placebo: orally daily
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib: 600 mg orally daily
  Other Names: Votrient
  Arms: Erlotinib + Pazopanib
Drug: Erlotinib — Erlotinib: 150 mg orally daily
  Other Names: Tarceva

SUMMARY:
This randomized, placebo-controlled, Phase II trial will compare the combination of erlotinib with pazopanib (providing concurrent EGFR and VEGFR inhibition) with erlotinib alone in the second- or third-line treatment of patients with advanced NSCLC. This study will be conducted though the Sarah Cannon Research Consortium, a community-based clinical trial network.

DETAILED DESCRIPTION:
Erlotinib is the current treatment standard for second- or third-line therapy of advanced NSCLC. Since angiogenesis inhibitors have also shown activity in NSCLC, the simultaneous inhibition of the EGFR and VEGF pathway may improve the efficacy of therapy. In a recently reported Phase III trial (Hainsworth et al. 2008), the combination of bevacizumab and erlotinib improved the Progression- Free-Survival (PFS) vs. erlotinib alone when given as second-line therapy in NSCLC (3.4 months vs. 1.7 months, respectively; HR 0.63). Pazopanib also inhibits the angiogenesis pathway, and may have advantages over bevacizumab including: (1) inhibition of other potentially important targets, including PDGFR; and (2) more convenient oral administration.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic confirmation of stage IIIB/IV NSCLC (squamous carcinoma, adenocarcinoma, or large cell carcinoma) per the American Joint Committee on Cancer Cancer Staging Manual, 6th edition. Patients with mixed tumors with small- cell elements are ineligible.
2. At least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques, or as >10 mm with spiral computerized tomography scan according to the Response Evaluation Criteria in Solid Tumors version 1.1 (Eisenhauer et al. 2009)
3. Failure of at least 1, and no more than 2, prior chemotherapy regimens for advanced disease (either due to progressive disease or toxicity).
4. Recovery from any toxic effects of prior therapy to ≤ grade 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
5. Completion of radiation therapy at least 28 days prior to the start of study treatment (not including palliative local radiation). Previously irradiated lesions in the advanced setting cannot be included as target lesions unless clear tumor progression has been observed since the end of radiation.
6. ECOG Performance Status of 0-2.
7. Adequate hematologic, hepatic and renal function.
8. A female is eligible to enter and participate in this study if she is of:

   * non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had hysterectomy, bilateral oophorectomy (ovariectomy), bilateral tubal ligation, is post-menopausal
   * childbearing potential, including any female who has had a negative serum pregnancy test within 1 week prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception.
9. Patients entering the study must be willing to provide a serum sample at baseline and at off-study for disease progression for correlative serum proteomic testing.
10. Willingness to provide a plasma sample at baseline, and at off-study for disease progression for correlative testing of circulating plasma biomarkers.
11. Patients entering this study must be willing to provide tissue from a previous tumor biopsy (if available) for correlative tissue testing.
12. Patients must be able to understand the nature of this study, give written informed consent, and comply with study requirements.

Exclusion Criteria:

1. Past or current history of neoplasm (other than the entry diagnosis), with the exception of treated non-melanoma skin cancer or carcinoma in-situ of the cervix, or other cancers cured by local therapy alone, and a disease-free survival ≥3 years.
2. Prior treatment with EGFR tyrosine kinase inhibitors or vascular endothelial factor receptor tyrosine kinase inhibitors for NSCLC. [Note: prior bevacizumab (Avastin®) use is permitted].
3. Prior use of an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
4. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by New York Heart Association classification
5. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 1 week prior to first dose of study drug. Screening with CNS imaging (CT or magnetic resonance imaging) is required only if clinically indicated or if the subject has a history of CNS metastases.
6. Women who are pregnant or lactating. All females of childbearing potential must have negative serum or urine pregnancy tests within 7 days prior to study treatment.
7. Poorly controlled hypertension [defined as systolic blood pressure of ≥150 mmHg or diastolic blood pressure of ≥90mmHg].
8. Presence of uncontrolled infection.
9. Prolongation of heart rate-corrected QT interval (QTc) ≥480 msec (using Bazett's formula).
10. Use of any of the medications on the prohibited medication list within 14 days of study treatment (with the exception of Amiodarone, which is prohibited from 6 months prior to screening through discontinuation from the study).
11. A serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
12. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
13. Minor surgical procedures (with the exception of the placement of portacath or other central venous access) performed less than 7 days prior to beginning protocol treatment.
14. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism (PE), or untreated DVT within the past 6 months.
15. Previous treatment with cetuximab.
16. Patients with hemoptysis or tumor cavitation at baseline.
17. Any prior history of hypertensive crisis or hypertensive encephalopathy.
18. Pulmonary hemorrhage/bleeding event within 6 weeks prior to beginning study treatment.
19. Any other non-pulmonary hemorrhage/bleeding event ≥ grade 3 within 28 days of study treatment.
20. Evidence or history of bleeding diathesis.
21. Serious non-healing wound, ulcer, or bone fracture.
22. Known or suspected allergy/hypersensitivity to any agent given in the course of this trial.
23. Clinically significant gastrointestinal (GI) abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (8):
- United States (8):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Suburban Hem Onc, Lawrenceville, Georgia
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collerville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib + Pazopanib | Erlotinib + Placebo
Started | 134 (One patient was enrolled but not treated) | 67
Completed | 0 (Patients remained on treatment until coming off for progression, toxicity or any other reason) | 0 (Patients remained on treatment until coming off for progression, toxicity or any other reason)
Not Completed | 134 | 67

BASELINE CHARACTERISTICS:
Population: All treated patients
Groups:
- Arm A: Erlotinib + Pazopanib
  Erlotinib: 150 mg orally daily
  Pazopanib: 600 mg orally daily
- Arm B: Erlotinib + Placebo
  Erlotinib: 150 mg orally daily
  Placebo: orally daily
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 134 | 67 | 201
Age, Continuous [Median (Full Range); unit: years] | 66 [35 to 88] | 67 [48 to 85] | 67 [35 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 28 | 91
  Male | 71 | 39 | 110
Region of Enrollment [Number; unit: participants] — Includes all treated patients
  participants
    United States | 134 | 67 | 201

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The length of time, in months, that patients were alive from first date of protocol treatment until worsening of disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 14 months
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 134 | 67
months | 2.6 [1.9 to 3.2] | 1.8 [1.7 to 2.0]

2. Secondary Outcome: Overall Survival
Description: The length of time, in months, that patients were alive from first date of protocol treatment until death.
Time Frame: 18 months
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 134 | 67
months | 6.76 [4.7 to 8.1] | 6.7 [5.0 to 9.3]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of patients having an objective benefit from treatment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 18 Months
Population: Includes all patients who were evaluated for response
Measure: Number; unit: percentage of evaluated participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 99 | 56
percentage of evaluated participants | 12.12 | 5.36

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 47/134 | 19/67
Other Adverse Events (participants affected / at risk) | 132/134 | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=134) | Arm B (N=67)
General disorders and administration site conditions - Other, disease progression (General disorders) | 8 | 4
Infections and infestations - Other, pneumonia (Infections and infestations) | 8 | 2
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Thromboembolic event (Vascular disorders) | 4 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 2 | 1
alanine aminotransferase increased (Investigations) | 2 | 0
aspartate aminotransferase increased (Investigations) | 2 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
blood bilirubin increased (Investigations) | 1 | 0
Cardiac disorders - Other, tachycardia (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
dizziness (Nervous system disorders) | 0 | 1
fever (General disorders) | 0 | 1
Gastrointestinal disorders - Other, hematemesis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, small bowel obstruction (Gastrointestinal disorders) | 1 | 0
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 1 | 0
hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other, bacteremia (Infections and infestations) | 1 | 0
Infections and infestations - Other, Staphylococcus (Infections and infestations) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Weight Loss (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=134) | Arm B (N=67)
Diarrhea (Gastrointestinal disorders) | 92 | 36
Fatigue (General disorders) | 68 | 30
Nausea (Gastrointestinal disorders) | 55 | 25
Anorexia (Metabolism and nutrition disorders) | 48 | 17
Proteinuria (Renal and urinary disorders) | 38 | 14
Rash (Skin and subcutaneous tissue disorders) | 34 | 16
Weight Loss (Investigations) | 36 | 11
Vomiting (Gastrointestinal disorders) | 32 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 | 12
Dehydration (Metabolism and nutrition disorders) | 27 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 10
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 27 | 6
Anemia (Blood and lymphatic system disorders) | 20 | 4
Platelet Count Decreased (Investigations) | 20 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 12 | 9
Rash Acneiform (Skin and subcutaneous tissue disorders) | 11 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 4
Dysgeusia (Nervous system disorders) | 14 | 3
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 14 | 1
Headache (Nervous system disorders) | 11 | 3
Dizziness (Nervous system disorders) | 10 | 3
Constipation (Gastrointestinal disorders) | 6 | 6
Mucositis (Gastrointestinal disorders) | 9 | 3
White Blood Cell Decreased (Investigations) | 11 | 1
Hypertension (Vascular disorders) | 9 | 2
Infections And Infestations - Other, Pneumonia (Infections and infestations) | 9 | 2
Fever (General disorders) | 7 | 3
General Disorders And Administration Site Conditions - Other, Disease Progression (General disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites